CLINICAL TRIAL: NCT03213197
Title: Feasibility of a Standardized Video for Patient Education and as a Decision Aid on Code Status for Patients in the Emergency Department Pending Admission to the Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Caitlin E. Loprinzi Brauer, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-009141
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Patient Education

STUDY DESIGN:
Intervention Model Description: Feasibility of a Standardized Video for Patient Education and as a Decision Aid on Code Status for Patients in the Emergency Department pending Admission to the Hospital
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPR video (Experimental): Patient watches a short CPR video
  Interventions: Other: CPR video

INTERVENTIONS:
Other: CPR video — Patient watches a short CPR video

SUMMARY:
The researchers hypothesize that patients and their families will be comfortable watching standardized CPR informational videos and that they would recommend that others watch the videos. Furthermore, the researchers hypothesize that patients and their families will find the videos helpful in their own end-of-life planning.

DETAILED DESCRIPTION:
The code status video, produced by experts in palliative medicine and end of life care, has been evaluated in a variety of healthcare settings to allow patients to make more informed decisions based on realistic information about resuscitation status. This video could be used as a supplement for clinical discussions and decision making. It is not meant to replace a careful, individualized discussion by the clinician with patients and their families, but appears to be a helpful tool to help educate patients in order for them to be better informed to make complicated decisions about their code status. The Emergency Department is an ideal setting to evaluate the video because they could improve patient understanding in an environment with inherently limited face-to-face provider time.

Specific Aims

1. To assess the satisfaction of patients and family members who view the video on cardiopulmonary resuscitation. This will be measured through use of a questionnaire asking them to score their comfort with watching the video and how likely they would be to recommend the video to others.
2. To assess if watching the standardized video changes patients' code status. This will be measured as what patients' code status was before and after watching the video.

ELIGIBILITY:
Inclusion Criteria

* Any patient in the Emergency Department whose disposition is listed as a full admission to the hospital
* Provider willingness to have patient watch the video and be available to answer questions after.
* Age > 65
* Ability to provide consent

Exclusion Criteria

* Does not speak English
* Hearing or visually impaired
* Prisoner or incarcerated
* Inability to provide consent according to attending Physician or Study Coordinator and legal power of attorney is not present

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Satisfaction of patients and family members in watching videos of cardiopulmonary resuscitation | 1 year
  This will be measured through use of a questionnaire asking them to score their comfort with watching the video and how likely they would be to recommend the video to others.

SECONDARY OUTCOMES:
The number of patients/families who will feel that the video was helpful in the decision regarding code status | 1 year
  To assess if watching the standardized video changes patients' code status. This will be measured as what patients' code status was before and after watching the video.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin E Loprinzi Brauer, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Not being shared....